CLINICAL TRIAL: NCT06758518
Title: Are Anxiety and Depressive Disorders Related to Carpal Tunnel Syndrome in Medical Students?
Brief Title: Study of the Carpal Tunnel Syndrome in Relation to Stress and Depression Among Medical Students
Acronym: CRS
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, AIKATERINI MARINI, MD, PhD, Researcher, University of Ioannina
Other Study IDs: 48955/17-12-2024
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-01

CONDITIONS: Carpal Tunnel Syndrome (CTS)
Keywords: carpal tunnel syndrome; anxiety; depression; medical students
MeSH Terms: conditions — Carpal Tunnel Syndrome; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- With carpal tunnel syndrome: Subjects with medial nerve disorders (clinical or ultrasound surface of the nerve over 12mm2).
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — there will be no intervention
  Other Names: no intervention

SUMMARY:
Participants will undertake validation of the median nerve and their anxiety and depression levels. Possible correlation will be searched.

DETAILED DESCRIPTION:
Medical students of the University of Ioannina will be submitted to ultrasound of the medial nerve as to assess its surface. Those with pathological findings will undertake a non-interventional electromyography test. Afterwards they will complete anonymously two validated tests regarding depression and anxiety (Yung ans STAI scales). Statistical analysis will be conducted with the question of correlation between median nerve dysfunction and psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* medical students

Exclusion Criteria:

* known pathology of the carpal joint

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: medical students of the university of ioannina
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Correlation of median nerve disorder with anxiety and/or depression | 1 month
  the measurement of the median nerve surface will be examined for correlation with depression or anxiety through self- questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School, University of Ioannina, Ioannina, Epirus, Greece

IPD SHARING:
Plan to Share IPD: No
No personal data of the students will be announced. All the study will be completed anonymoously.